CLINICAL TRIAL: NCT04738383
Title: Feasibility and Acceptance of Changes in Medical Supervision of Exercise Groups in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: National Paralympic Committee Germany (NPCG) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-28-MB
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Rehabilitation; Rehabilitation Exercise; Organization and Administration; Feasibility Studies
Keywords: perceived safety; cardiac rehabilitation; exercise; medical supervision
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: control group and 3 different forms of medical supervision
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Version 1: Paramedic (Experimental): Physician is replaced by a paramedic, but the physician still acts as a supervisor.
  Interventions: Procedure: Version 1: Paramedic
- Version 2: Physician-on-call (Experimental): Physician is not present, but is on call.
  Interventions: Procedure: Version 2: Physician-on-call
- Version 3: Trained instructor (Experimental): Physician acts as a supervisor, but is not constantly present. The instructor received a special training preparing for emergency cases.
  Interventions: Procedure: Version 3: Trained instructor
- Control group (No Intervention): The sessions take place in the usual way, meaning that a physician is present in every session.

INTERVENTIONS:
Procedure: Version 1: Paramedic — Instead of a physician, who is constantly present, a paramedic is present next to the instructor during the sessions, who can give first aid in case of an emergency and bridge the time until the ambulance arrives on site. The physician still acts as a supervisor visiting the group roughly every six weeks.
  Arms: Version 1: Paramedic
Procedure: Version 2: Physician-on-call — This version implicates that a physician is not physically present but is on call during the sessions and must be constantly accessible by phone and able to arrive within three minutes in case of an emergency. To ensure this, version two should be implemented in facilities, which are linked to cardiac or rehabilitation center.
  Arms: Version 2: Physician-on-call
Procedure: Version 3: Trained instructor — The sessions take place with the instructor only, who receives a comprehensive emergency training before and during the model phase and replaces the constantly present physician. Just like in the previous versions the physician still acts as a supervisor visiting the group roughly every six weeks.
  Arms: Version 3: Trained instructor

SUMMARY:
Exercise groups are a form of rehabilitation sport that is offered to cardiac patients (e.g. after a heart attack) in long-term rehabilitation. In Germany, the constant presence of a physician is mandatory. In order to meet the increasing demand for heart groups, the present study implements emergency care during the heart group sessions with three alternatives: paramedics, physician-on-call or specially trained instructors.

In the present study the investigators compare these alternatives (three experimental conditions) with the conventional way (control condition). Perceived safety, trust, acceptance and organisational feasibility are the main outcomes of the study. The methods used are questionnaires to the participants, instructors, organizers and, if applicable, paramedics. Additionally, partially structured interviews with attending physicians are conducted according to an interview guide.

DETAILED DESCRIPTION:
Exercise groups are a form of rehabilitation sport that is offered to cardiac patients (e.g. after a heart attack) in long-term rehabilitation. In Germany it is paid for by the health insurance, when certain quality criteria are fulfilled. Among others, the constant presence of a physician is mandatory. In order to meet the increasing demand for heart groups, the National Paralympic Committee Germany (NPCG) received a special permit to try other forms of medical care during a pilot project. In this so-called "supervisor conception" the physician focuses on higher-level supervision for several exercise groups. Emergency care during the heart group sessions is ensured with three alternatives: by paramedics, by a physician-on-call or by specially trained instructors.

In the present study the investigators compare these alternatives (three experimental conditions) with the conventional way (control condition). Before the start of the research project, the different versions were defined and approved by the NPCG and other responsible actors in German rehabilitation sport. The project is implemented for 12 months.

The objectives of the evaluation are:

* Safety and acceptance of the participants, instructors and supervisors with regard to medical care, consultation and cooperation, feasibility and communication between the interfaces.
* Learning effects and implementation of the training measures for emergency management and health education measures
* Implementability of the supervisor conception in the clubs and regional associations of the three model regions and transferability on the clubs and state associations of the NPCG.

The methods used are questionnaires to the participants, instructors, organizers and, if applicable, paramedics, in which the assessment of the respondents is measured for perceived safety, acceptance and feasibility. The questionnaires to the participants and instructors are carried out during a session by employees of the participating sports clubs. The organizers fill out their questionnaires at a self-chosen time point. The questionnaires were developed by the university and were sent out after the client has given his/her informed consent.

Additionally, partially structured interviews with attending physicians are conducted according to an interview guide. The questions address the physicians' assessment of safety, acceptance and feasibility of the supervisor conception.The guidelines are developed by us and are used by us after approval by the client. We conduct the interviews ourselves by telephone and evaluate them.

ELIGIBILITY:
Inclusion Criteria:

* For participants: Participation in the heart sports group with the consent of the prescribing physician

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Trust at M3 | Month 3 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Trust of the participants, instructors, organizers and paramedics towards the three alternative versions in cardiac rehabilitation. It is measured with one question offering a six-point Likert scale. The feasibility criterion is met, if 50% or less of the respondents tick box 5 or 6 (strong rejection/ no trust).
Trust at M10 | Month 10 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Trust of the participants, instructors, organizers and paramedics towards the three alternative versions in cardiac rehabilitation. It is measured with one question offering a six-point Likert scale. The feasibility criterion is met, if 50% or less of the respondents tick box 5 or 6 (strong rejection/ no trust).
Willingness at M3 | Month 3 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Willingness of the participants, instructors and organizers to implement the versions of the supervisor conception. It is assessed with a "yes-no-question" in the questionnaire. The feasibility criterion is met, if 50% or less of the respondents answer "no".
Willingness at M10 | Month 10 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Willingness of the participants, instructors and organizers to implement the versions of the supervisor conception. It is assessed with a "yes-no-question" in the questionnaire. The feasibility criterion is met, if 50% or less of the respondents answer "no".
Potential at M3 | Month 3 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Assessment of the organizers, instructors and paramedics if the supervisor conception has the potential to be able to offer more cardiac rehabilitation groups. It is measured with one question offering a six-point Likert scale. The feasibility criterion is met, if 50% or less of the respondents tick box 5 or 6 (strong rejection/ no potential).
Potential at M10 | Month 10 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Assessment of the organizers, instructors and paramedics if the supervisor conception has the potential to be able to offer more cardiac rehabilitation groups. It is measured with one question offering a six-point Likert scale. The feasibility criterion is met, if 50% or less of the respondents tick box 5 or 6 (strong rejection/ no potential).
Costs at M3 | Month 3 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Organizers are asked if the supervisor conception causes more, less or the same amount of costs compared to the conventional cardiac rehabilitation group. It is measured with one question offering a seven-point Likert scale. The feasibility criterion is met, if 50% or less of the respondents tick box 6 or 7 (more or much more costs).
Costs at M10 | Month 10 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  Organizers are asked if the supervisor conception causes more, less or the same amount of costs compared to the conventional cardiac rehabilitation group. It is measured with one question offering a seven-point Likert scale. The feasibility criterion is met, if 50% or less of the respondents tick box 6 or 7 (more or much more costs).

OTHER OUTCOMES:
Other questions on the implementation of the concept (M3) | Month 3 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  The questionnaire containing the 4 primary outcome questions includes also other questions on the implementation of the concept, e.g. the supervision, the communication between actors and the activity of the exercise instructor. No score is calculated.
Other questions on the implementation of the concept (M10) | Month 10 of the intervention. The clubs received the questionnaires by mail and had one month to fill them out and send them back.
  The questionnaire containing the 4 primary outcome questions includes also other questions on the implementation of the concept, e.g. the supervision, the communication between actors and the activity of the exercise instructor. No score is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Ewald, Study Director — National Paralympic Committee Germany (NPCG); Michael Brach, Prof. Dr., Principal Investigator — Universität Münster
Locations (4):
- Germany (4):
  - Behinderten-Sportverband Niedersachsen e.V., Hanover, Lower Saxony
  - National Paralympic Committee Germany (NPCG), Frechen, North-Rhine Westfalia
  - Instiute of Sport and Exercise Sciences, Münster, North-Rhine Westfalia
  - Sächsischer Behinderten- und Rehabilitationssportverband e. V., Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No